CLINICAL TRIAL: NCT06771713
Title: Brief Pain Reprocessing Therapy: An Optimized Integrative Exposure Intervention for Veterans With Chronic Low Back Pain
Brief Title: Brief Pain Reprocessing Therapy in Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Sturgeon, Clinical Assistant Professor of Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00255952; GRANT14011002 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lower Back Pain (CLBP)
Keywords: Veterans; Telehealth based intervention; Brief Pain Reprocessing Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Pain Reprocessing Therapy (BPRT) (Experimental): Participants will have therapy over the internet.
  Interventions: Behavioral: Brief Pain Reprocessing Therapy (BPRT)

INTERVENTIONS:
Behavioral: Brief Pain Reprocessing Therapy (BPRT) — Participants will have three 90-minute behavioral intervention sessions over a 3-week period, completing 35 days of brief daily assessments, and one additional set of questionnaires.
  Participants will also complete study questionnaires at 1, 2, 3, and 6 months after attending the 3 behavioral intervention sessions.

SUMMARY:
This research is studying whether a Zoom-based behavioral intervention may have an impact as a treatment for Veterans with Chronic Low Back Pain (CLBP).

The study will examine:

* The acceptability of the Brief Pain Reprocessing Therapy (BPRT) intervention
* The feasibility of the BPRT intervention
* The safety of the BPRT intervention

DETAILED DESCRIPTION:
This study will take place remotely and there will be no on-site visits.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain that has lasted greater than 6 months, with pain on at least half of these days
* Must provide verification of being an Armed Service Veteran.
* Able to read, write and speak English
* Internet access and audio-conferencing capability (e.g., Zoom meetings by phone or computer) in the home

Exclusion Criteria:

* Self-reported evidence of a separate medical condition (e.g., rheumatoid arthritis), acute injury in the past 12 months (e.g., self-reported spinal fracture), self-reported loss of bowel or bladder control in the past year (which may indicate presence of cauda equina syndrome), or evidence of presence of a metastasizing cancer requiring treatment
* Pending surgical procedures or interventional therapies (e.g., spinal injections) within the next 12 months
* Confirmed/suspected pregnancy
* Evidence of other conditions that may preclude participants from understanding or being able to participate in study procedure (e.g., schizoaffective disorder, suspected or diagnosed dementia)
* Currently receiving cognitive-behavioral therapy or other psychological therapies for pain
* Open litigation in the past 1 year, as assessed in preliminary study screening.
* Any other diseases or conditions that would make a patient unsuitable for study participation as determined by the site principal investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of and satisfaction with treatment base on the mean scores on the Treatment Evaluation Inventory (TEI-SF) assessed at T5 (approximately day 35) | Approximately day 35 (post treatment)
  The TEI-SF is a validated instrument for behavioral interventions. There are 9 questions that participants answer from 1 (strongly disagree) - 5 (strongly agree) with a range of (9-45) with a higher score indicating greater acceptability. Scores at 27 or above will denote moderate acceptability of the intervention.
Feasibility will be accessed by participant adherence | Up to approximately day 35 (post treatment)
  Adherence to the intervention will be determined by at least 80% attendance of intervention sessions, completion of daily assessment, and self-reported adherence to home-base exposure practices, completion of pre/post session and pre/post interventions.
Feasibility will be accessed by feedback from the Qualitative Interviews | Approximately day 35 (post treatment)
  Qualitative Interviews will occur after conclusion of the intervention period to address areas of improvement in future iterations of the intervention.
Safety will be assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS 29) pain intensity | Baseline, up to day 35 post treatment
  There is 1 question that participants will answer pain level from 0 (not at all) - 10 (worst pain imaginable).
Safety will be assessed by the PROMIS Depression scale | Baseline, up to day 35 post treatment
  Participants will answer 4 questions 1 (never) -5 (always). There is a range of scores from 4-20 with a higher score indicating higher levels of depression.
Safety will be assessed by the PROMIS Anxiety scale | Baseline, up to day 35 post treatment
  Participants will answer 4 questions 1 (never) -5 (always). There is a range of scores from 4-20 with a higher score indicating higher levels of anxiety.
Safety will be assessed by the Patient Global Impression of Change (PGIC) | Baseline, up to day 35 post treatment
  There is 1 question that participants will select from 1 (very much improved) - 7 (very much worse).
Safety assessed by the number of Adverse events and Serious adverse events T6 (Day 60) - T9 (Day 210) | T6 (Day 60) - T9 (Day 210)
  Adverse events will be classified as serious or non-serious (per protocol). These will be assessed by items such as death, life-threatening event, hospitalization, emergency room visits, persistent or significant disability/incapacity, suicide plans or attempts.

SECONDARY OUTCOMES:
Change from T1 (day 1) to T6 (Day 60) in Tampa Scale of Kinesiophobia (TSK) | T1 (Day 1) - T6 (Day 60)
  There are 17 questions that participants will select from a score of 1 (strongly disagree) - 4 (strongly agree). A total score is calculated after reversing items 4, 8, 12 and 16. The scores range between 17-68. A high score on the scale indicates that the person has a high level of kinesiophobia.
Change from T1 to T6 (Day 60) pain intensity | T1 (Day 1) - T6 (Day 60)
  There is 1 question that participants will answer pain level from 0 (not at all) - 10 (worst pain imaginable).
Change from T1 to T6 (Day 60) PROMIS Pain Interference | T1 (Day1) - T6 (Day 60)
  Participants will answer 4 questions 1 (not at all) -5 (very much). There is a range of scores from 4-20 with a higher score indicating higher levels of interference.

CONTACTS AND LOCATIONS:
Overall Officials: John Sturgeon, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No